CLINICAL TRIAL: NCT06545669
Title: C-Raven: Pilot Randomized Controlled Trial (RCT) of an Avatar-delivered Computerized Intervention for Tobacco Cessation With Community Health Worker Linkage to Lung Cancer Screening in Baltimore City
Brief Title: C-Raven, a Virtual Tobacco Cessation Intervention in the Community
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government); Walgreens (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00450397
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Community Health Workers

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomly assigned to intervention or no intervention. Outcomes for those who receive the intervention will be compared to outcomes for those who do not receive the intervention. Those who do not receive the intervention during the initial study period will receive it at the end, to ensure access to treatment for all participants.
Masking Description: The statistical analyst will not be made aware of which treatment group received the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- C-Raven + CHW Smoking Cessation Intervention (Experimental): Participants will receive a virtual counselor intervention for smoking cessation, be offered the opportunity to utilize nicotine replacement therapies, participate in shared decision-making around lung cancer screening, and be supported by a community health worker. Participants will be followed for a total of 6 months. Assessments will be conducted at baseline, 1 month, 3 months, and 6 months.
  Interventions: Behavioral: C-Raven Virtual Tobacco Cessation Counseling; Drug: Nicotine Replacement Product; Other: Community Health Worker; Other: Lung Cancer Screening
- No Intervention (No Intervention): Participants will not receive any intervention during the first 6 months of the study. The participants will receive the study intervention at the end of 6 months, to ensure access to treatment for all participants.

INTERVENTIONS:
Behavioral: C-Raven Virtual Tobacco Cessation Counseling — A two-module tobacco cessation intervention that involves interaction with a virtual counselor and includes instruction about addiction and the use of pharmacotherapy for cessation. Each module takes approximately 20 minutes to complete.
  Arms: C-Raven + CHW Smoking Cessation Intervention
Drug: Nicotine Replacement Product — Participants will be offered a 12-week supply of nicotine patches and either nicotine gum or lozenges.
  Arms: C-Raven + CHW Smoking Cessation Intervention
Other: Community Health Worker — A community health worker will meet with each participant throughout the study period to teach appropriate NRT usage, discuss barriers/facilitators to NRT use and cessation, conduct shared decision-making about lung cancer screening, and provide health system navigation when needed.
  Arms: C-Raven + CHW Smoking Cessation Intervention
Other: Lung Cancer Screening — After participating in shared decision-making, eligible participants will be referred to their primary care physician or existing specialist to complete lung cancer screening.
  Arms: C-Raven + CHW Smoking Cessation Intervention

SUMMARY:
In low-income housing units in Baltimore, the investigators propose to conduct a pilot two-arm hybrid type 1 effectiveness-implementation RCT comparing a) an avatar-delivered computerized intervention (CI) for tobacco cessation augmented with CHW support and navigation to lung cancer screening to b) a waitlist control.

With a sample of participants from public housing units (N=30), the investigators will collect data on feasibility of recruitment, intervention engagement and completion, and short-term smoking cessation outcomes. Individuals will be assessed at baseline, 1 month, 3 months, and 6 months. At the 3-month time point, the investigators will conduct interviews with a subset of pilot participants to collect qualitative data on intervention acceptability.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized controlled trial of an avatar-delivered computerized intervention for tobacco cessation and CHW support to collect data on the feasibility of recruitment, intervention engagement and completion, and short-term smoking cessation outcomes. Individuals will be assessed at baseline, one month, three months, and six months. At the end of three months, the investigators will conduct follow-up interviews with a subset of pilot participants to collect qualitative data on intervention acceptability. Based on the information collected in these efforts, the investigators will make iterative improvements to the existing intervention, aligned with user-experience design procedures.

Participants (N=30) will be recruited through flyers posted in and around the housing units and distributed to tenants by housing unit staff. Flyers will describe the study and contain a study phone number to call. Information may also be distributed by study staff during non-study-related health and wellness activities conducted at the sites. At initial contact, a study staff member will discuss the study purpose and determine eligibility. If eligible, the staff member will proceed to discuss requirements, review risks and benefits, and obtain informed consent from interested participants.

Consent process: After confirming eligibility with screening questions via phone, potential participants will be offered the option of reviewing the study information and consent form over a Zoom video conference. Regardless of whether the participants choose to review this information in advance, all potential participants will complete the consent process and sign the consent form at the beginning of the first in-person visit, which will be conducted on-site at the participants housing community.

Randomization: Following consent, participants will be randomized to the intervention group or a control group. The control group will not receive any intervention during the first 6 months of the study, but at the end of 6 months will receive the full computer intervention and abbreviated CHW support to ensure access to treatment for all participants.

Baseline Assessment: This will occur on the same day as the in-person portion of the consent process. Initial evaluation will comprise a number of questionnaires/assessments, including demographics, a clinical history, a tobacco use history, and a number of tobacco-related measures. Assessments will be self-administered via tablet computer.

Intervention:

Computer-Delivered Intervention (CDI) Session 1: Following the baseline assessment, participants will receive computer-delivered counseling via a study-provided iPad delivered in a private room. The CDI consists of 1) a menu-driven, web-based intervention that is delivered by a virtual counselor. The intervention takes 20 minutes to complete. At the conclusion of session 1, the participant will be offered nicotine patches provided by the study (1 month supply, remainder given at follow-up visits). The initial dosing of the nicotine patches will be determined based on cigarettes consumed per day (>10: 21mg patch, 5-10: 14mg patch, <5: 7mg patch). If there is any question regarding eligibility or appropriate dosing, the CHW will consult with a study physician. With the CHW, the participant will learn correct application, and will monitor the participants nicotine replacement therapy (NRT) experience in discussion with the CHW.

Computer-Delivered Intervention (CDI) Session 2: Session 2, delivered approximately one week later, focuses on the cycle of addiction and use of pharmacotherapy (e.g., NRT, bupropion, varenicline). This intervention also takes about 20 minutes to complete. At the conclusion of session 2, the participant will be offered nicotine gum or lozenges provided by the study (1 month supply, remainder given at follow-up visits). This session also includes an in-session experience of using NRT gum or lozenge, with CHW guidance to ensure correct use.

Community Health Workers (CHWs): A CHW will meet with each participant for both Sessions 1 and 2 and will do the following: 1) Teach appropriate NRT use technique as above, 2) Follow up with patients remotely via phone or video conference whenever possible, up to twice weekly for 12 weeks (4 weeks for control group receiving delayed intervention), to discuss barriers/facilitators to maintenance of NRT use and tobacco cessation; 3) Review a video and decision-making guide for lung cancer screening and provide linkage to lung cancer screening if the participant is eligible and interested, including linkage to insurance enrollment assistance, if needed; 4) For individuals requiring follow up for positive findings on lung CT, work with participants to navigate the process; 5) Link interested participants to the QuitLine; 6) At the end of the study, link to medical providers for additional tobacco cessation therapy if participant interested (e.g., varenicline, bupropion).

Linkage to Lung Cancer Screening: Participants eligible for and interested in CT Lung cancer screening (age ≥50, ≥20 pack year smoking history) will be referred to the participants primary care physician (PCP) or existing specialist for further discussion and ordering. The CTs are optional and will not be provided as part of the research study. The CHW will assist with linking patients without a PCP or existing specialist with resources to establish care. For participants who choose to proceed with screening, the investigators will request the results of the CT scan to track completion and general result category (Normal/Normal with Minor Findings/Abnormal Needing Short-Term Follow-Up/Abnormal Needing Immediate Follow-Up).

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older Current tobacco use with >100 cigarettes smoked in their lifetime
* English speaking (intervention currently in English only and housing units are in largely English-speaking neighborhoods)
* Considering smoking cessation
* Planning to remain in current housing unit for 9 months

Exclusion Criteria:

* Current use of pharmacological treatment for tobacco cessation
* Contraindication to nicotine replacement therapy
* Current engagement in formal smoking cessation program
* Major cognitive or psychiatric impairment
* Severe hearing impairment
* Investigator discretion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Acceptability and Feasibility as assessed by number of barriers | 1 month, 3 months, 6 months
  Acceptability and Feasibility will be assessed through quantitative and qualitative data on factors including (e.g., number of participant engagement, number of barriers,completion of modules, number of sessions with CHW).
Acceptability and Feasibility as assessed by completion of modules | 1 month, 3 months, 6 months
  Acceptability and Feasibility will be assessed through quantitative and qualitative data on factors including (e.g., number of participant engagement, number of barriers,completion of modules, number of sessions with CHW).
Acceptability and Feasibility as assessed by number of sessions with CHW | 1 month, 3 months, 6 months
  Acceptability and Feasibility will be assessed through quantitative and qualitative data on factors including (e.g., number of participant engagement, number of barriers,completion of modules, number of sessions with CHW).

SECONDARY OUTCOMES:
Readiness to quit smoking as assessed by The Readiness Ruler | 1 month, 3 months, 6 months
  The Readiness Ruler is a brief measure of motivation, which prompts patients with a 10-point visual analog scale on which the participant rates readiness, with a score of 0 reflecting "not ready," and a score of 10 reflecting "ready."
Number of participants that start nicotine replacement therapy uptake | 1 month, 3 months, 6 months
  Number of participants that start using NRTs at any point during the study period
Number of participants that continue use of nicotine replacement therapy | 1 month, 3 months, 6 months
  Number of participants that continue to use NRTs
Number of participants that attempt to quit | 1 month, 3 months, 6 months
  Number of participants that attempt to quit
Number of quit attempts | 1 month, 3 months, 6 months
  Number of quit attempts each participants makes during the study period
Number of participants that maintain cessation | 1 month, 3 months, 6 months
  Number of participants that have maintained cessation for at least one week prior to the assessment
Number of participants that utilize Quit Line services | 1 month, 3 months, 6 months
  Number of participants that chose to utilize Quit Line services at any point during the study
Number and frequency of interactions with the community health worker | 1 month, 3 months, 6 months
  Engagement with community health worker
Participant satisfaction as assessed by the C-Raven Satisfaction Scale | 1 month, 3 months, 6 months
  Overall satisfaction with the intervention. This will be measured with a 21-item questionnaire which uses a 5-item Likert Scale for each question (range 21-105). Higher scores indicate greater satisfaction. Answers of "agree" and "strongly agree" will be evaluated across the intervention components.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Ellison-Barnes, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No